CLINICAL TRIAL: NCT06476080
Title: Ultrasound Guided Serratus Anterior Versus Erector Spinae Block in Pain Alleviation in Acute Herpes Zoster: A Prospective Comparative Study
Brief Title: Ultrasound Guided Serratus Anterior Versus Erector Spinae Block in Pain Alleviation in Acute Herpes Zoster
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Ass professor anesthesia and pain, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1084
Record Dates: First submitted 2024-06-15; First posted 2024-06-26 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Acute Herpes Zoster Neuropathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): 800 mg acyclovir, 5 times / day, orally administered, for one week, acetaminophen 1000 mg per day, topical calamine lotion)
- Erector spinae group (Active Comparator): 800 mg acyclovir, 5 times / day, orally administered, for one week, acetaminophen 1000 mg per day, topical calamine lotion)+ 25 ml bupivacaine 0.25% plus 8 mg dexamethasone
  Interventions: Procedure: ultrasound guided erector spine block
- Serratus anterior group (Active Comparator): 800 mg acyclovir, 5 times / day, orally administered, for one week, acetaminophen 1000 mg per day, topical calamine lotion)+ 25 ml bupivacaine 0.25% plus 8 mg dexamethasone
  Interventions: Procedure: Serratus anterior block

INTERVENTIONS:
Procedure: ultrasound guided erector spine block — Ultrasound guided thoracic erector spinae block
  Arms: Erector spinae group
Procedure: Serratus anterior block — Ultrasound guided serratus anterior block
  Arms: Serratus anterior group

SUMMARY:
Acute herpes zoster pain is very severe . Conventional analgesics may be of no value. Regional blocks may play a role

ELIGIBILITY:
Inclusion Criteria:

* Adult population between 30 and 75 years old.
* Unilateral painful thoracic herpetic eruption of less than one week duration.
* VAS more than or equal 4, persistent pain in spite of proper antiviral and analgesic therapy, (800 mg oral acyclovir, 5 times per day, for one week), pregabalin 300 mg per day, acetaminophen 1000 mg per day, topical calamine lotion).

Exclusion Criteria:

* Diabetic patients.
* Painful herpetic eruptive vesicles more than one week.
* Abdominal herpetic eruptions.
* Non-compliant on anti-viral (bulbar palsy for example).
* Co-malignancy or radiotherapy.
* Steroid therapy > 5 mg prednisolone or its equivalent.
* Infections or hematoma at site of injection.
* Coagulopathy (chronic kidney or liver disease, clopidogrel use).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
pain score | immediate after injection, 1 week, 1, 3 months
  Visual analogue scale from 0 to 10. 0= NO pain, 1-3=mild tolerable pain, 4-6= moderate pain, 7-10= severe untearable pain.

SECONDARY OUTCOMES:
Number of patients with pain recurrence | 1 week, 1, and 3 months
  Number of patients in need for re-injection
analgesic consumption | 1 week, 1, and 3 months
  total amount dose of analgesics used
Incidence of treatment related adverse events | immediately after injection
  hypotension, bradyarrhythmia, hematoma